CLINICAL TRIAL: NCT06733233
Title: A Multicenter, Prospective Phase II Single-arm Study Evaluating the Efficacy and Safety of Neoadjuvant Treatment with T-DXd in Combination with an Immune Checkpoint Inhibitor in HR-positive HER2 Low-expressing Chinese Patients with Early-stage Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of De Trastuzumab (T-DXd) in Combination with Immunotherapy for the Neoadjuvant Treatment of HR-positive HER2 Low-expressing Chinese Patients with Early-stage Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Huijin Wang, Director of Thyroid and Breast Disease Center, Guangzhou Women and Children's Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 158A01
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer, Estrogen Receptor-Positive; HER2 Low Breast Cancer
Keywords: Breast cancer; immunotherapy; DS8201; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Subjects who are eligible for the study and have signed informed consent will receive T-DXd in combination with an immune checkpoint inhibitor. The specific dosing regimen is as follows: T-DXd (5.4 mg/kg i.v. q3w) every 3 weeks for a total of 8 courses. Teraplizumab (240 mg/kg i.v. q3w), 1 course every 3 weeks for a total of 8 courses. Upon discontinuation of the study, subjects will receive post-neoadjuvant therapy according to local clinical criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- T-DXd combined with immune checkpoint inhibitor (Experimental)
  Interventions: Drug: T-DXd combined with immune checkpoint inhibitor

INTERVENTIONS:
Drug: T-DXd combined with immune checkpoint inhibitor — Subjects who are eligible for the study and have signed informed consent will receive T-DXd in combination with an immune checkpoint inhibitor. The specific dosing regimen is as follows: T-DXd (5.4 mg/kg i.v. q3w) every 3 weeks for a total of 8 courses. Teraplizumab (240 mg/kg i.v. q3w), 1 course every 3 weeks for a total of 8 courses.

SUMMARY:
This is a prospective, open-label, multicenter, single-arm clinical study designed to compare the efficacy and safety of neoadjuvant treatment with T-DXd in combination with an immune checkpoint inhibitor in patients with primary intermediate- to high-risk HR-positive, HER2-overexpressing early-stage breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant therapy, a systemic therapy administered prior to localized treatments such as surgery, has become a key component in the management of non-metastatic breast cancer. Neoadjuvant chemotherapy is often used to treat early-stage, high-risk hormone receptor-positive (HR+) breast cancer; however, the rate of pathological complete remission(pCR) is only 5-8 %. Moreover, neoadjuvant chemotherapy has significant toxicity, with approximately 25-40% of patients discontinuing chemotherapy or reducing their dosage due to side effect.

Much evidence suggests that immune checkpoint inhibitors (ICIs) combined with chemotherapy significantly increase pCR rates in HR+ breast cancer.

The CheckMate 7FL study evaluated the efficacy of ICI (nabulizumab) in early-stage HR-positive breast cancer, and ICI in combination with chemotherapy increased the pCR rate to 24%, compared to 13.8% in the chemotherapy arm[4].

The Keynote756 clinical trial demonstrated for the first time that the addition of an ICI (pembrolizumab) to a neoadjuvant chemotherapy regimen for early-stage, high-risk ER+/HER2- breast cancer significantly increased patients' pCR rates. These clinical trials imply that ICIs in combination with chemotherapy can provide more benefit to patients with early-stage breast cancer compared to traditional neoadjuvant chemotherapy treatments.

Trastuzumab deruxtecan (DS-8201a, T-DXd) is a novel HER2-targeted antibody-drug coupling (ADC) approved by the FDA and NMPA for the treatment of HER2-positive and HER2-low expressing metastatic breast cancer.

The BEGONIA study showed that Dato-DXd in combination with ICI (doxorubicinumab) for advanced triple-negative breast cancer had an ORR of up to 79%, which is superior to the efficacy of current ICIs in combination with chemotherapy; The DS8201-A-U105 study evaluated the efficacy of T-DXd in combination with navulizumab in HER2+ and HER2-low advanced breast cancer, with an ORR of 65.6% in the HER2+ and 50% in the HER2-low-expressing population, and the combination of T-DXd with navulizumab did not increase any overall toxicity.

The TALENT study explored the efficacy of T-DXd neoadjuvant therapy in patients with HR-positive HER2 low-expression early breast cancer. The results showed that T-DXd alone or in combination with ET achieved promising efficacy, with an ORR of 68% and a CR of 8% for T-DXd alone, indicating that T-DXd can also demonstrate very significant anti-tumor effects in early-stage breast cancer.

In view of the impressive efficacy and manageable safety of T-DXd in combination with ICIs in breast cancer patients, we designed this investigator-initiated clinical study with intermediate- and high-risk HR-positive HER2 low-expressing early-stage breast cancer patients to evaluate the efficacy and safety of T-DXd in combination with ICIs in early-stage HR-positive HER2 low-expressing breast cancer patients in a Chinese population.

This is a prospective, open-label, multicenter, single-arm clinical study designed to compare the efficacy and safety of neoadjuvant treatment with T-DXd in combination with an immune checkpoint inhibitor in patients with primary intermediate- to high-risk HR-positive, HER2-overexpressing early-stage breast cancer. Subjects who are eligible for the study and have signed informed consent will receive T-DXd in combination with an immunosuppressant. The specific dosing regimen is as follows:

T-DXd (5.4 mg/kg i.v. q3w) every 3 weeks for a total of 8 courses. Teraplizumab (240 mg/kg i.v. q3w), 1 course of treatment every 3 weeks for a total of 8 courses of treatment Upon discontinuation of the study, subjects will receive post-neoadjuvant therapy according to local clinical criteria.

Subjects will end study treatment if disease progression, intolerable toxicity, withdrawal of informed consent, or discontinuation of dosing is necessary in the judgment of the investigator occurs during the study treatment period, after which they will continue to receive follow-up, including metastatic disease recurrence and safety follow-up.

Subjects who complete surgical treatment will be followed for at least 3 years for the study endpoints of event-free survival (EFS), invasive disease-free survival (IDFS), overall survival (OS), and safety assessment. Safety data will be collected from the time of signing the informed consent form until 28 days after the end of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 18 and 70 at the time of signing the informed consent form.
2. An Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
3. Previously untreated, operable invasive breast cancer measuring greater than 2.0 centimeters (cT2) with positive clinical lymph nodes (cN1/cN2); or clinically staged T3-T4, clinically lymph node-negative (N0) or clinically lymph node-positive (cN1/cN2) without distal metastases.
4. Tumors with low levels of HER2 expression by immunohistochemistry (IHC), defined as IHC 1+ or IHC 2+ and FISH negative.
5. Tumor documented as HR-positive (ER and/or PgR-positive [ER or PgR ≥1%] by local assessment according to ASCO-CAP guidelines).
6. Patients who agree to undergo surgical treatment for breast cancer when they meet surgical criteria after neoadjuvant therapy.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer and bilateral breast cancer
2. Previous history of invasive breast cancer.
3. Previous history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS)
4. Other malignant tumors within 5 years, excluding cured carcinoma in situ of the cervix and non-melanoma skin cancers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete remission | 3 years

SECONDARY OUTCOMES:
event free survival | 3 years
invasive disease free survival | 3 years
overall survival | 3 years

OTHER OUTCOMES:
dose-limiting toxicities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Jie director, Doctor, Principal Investigator — Women and Children's Medical Center of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: Yes
Disease information of participants, Evaluation of treatment outcomes for participants
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025-01-01 to 2030-01-01

REFERENCES:
- [Background] Martin M, Pandiella A, Vargas-Castrillon E, Diaz-Rodriguez E, Iglesias-Hernangomez T, Martinez Cano C, Fernandez-Cuesta I, Winkow E, Perello MF. Trastuzumab deruxtecan in breast cancer. Crit Rev Oncol Hematol. 2024 Jun;198:104355. doi: 10.1016/j.critrevonc.2024.104355. Epub 2024 Apr 16. PMID 38621469
- [Background] Eskander RN, Sill MW, Beffa L, Moore RG, Hope JM, Musa FB, Mannel R, Shahin MS, Cantuaria GH, Girda E, Mathews C, Kavecansky J, Leath CA 3rd, Gien LT, Hinchcliff EM, Lele SB, Landrum LM, Backes F, O'Cearbhaill RE, Al Baghdadi T, Hill EK, Thaker PH, John VS, Welch S, Fader AN, Powell MA, Aghajanian C. Pembrolizumab plus Chemotherapy in Advanced Endometrial Cancer. N Engl J Med. 2023 Jun 8;388(23):2159-2170. doi: 10.1056/NEJMoa2302312. Epub 2023 Mar 27. PMID 36972022
- [Background] Spring LM, Gupta A, Reynolds KL, Gadd MA, Ellisen LW, Isakoff SJ, Moy B, Bardia A. Neoadjuvant Endocrine Therapy for Estrogen Receptor-Positive Breast Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1477-1486. doi: 10.1001/jamaoncol.2016.1897. PMID 27367583
- [Background] Tarantino P, Jin Q, Tayob N, Jeselsohn RM, Schnitt SJ, Vincuilla J, Parker T, Tyekucheva S, Li T, Lin NU, Hughes ME, Weiss AC, King TA, Mittendorf EA, Curigliano G, Tolaney SM. Prognostic and Biologic Significance of ERBB2-Low Expression in Early-Stage Breast Cancer. JAMA Oncol. 2022 Aug 1;8(8):1177-1183. doi: 10.1001/jamaoncol.2022.2286. PMID 35737367
- [Background] Denkert C, Seither F, Schneeweiss A, Link T, Blohmer JU, Just M, Wimberger P, Forberger A, Tesch H, Jackisch C, Schmatloch S, Reinisch M, Solomayer EF, Schmitt WD, Hanusch C, Fasching PA, Lubbe K, Solbach C, Huober J, Rhiem K, Marme F, Reimer T, Schmidt M, Sinn BV, Janni W, Stickeler E, Michel L, Stotzer O, Hahnen E, Furlanetto J, Seiler S, Nekljudova V, Untch M, Loibl S. Clinical and molecular characteristics of HER2-low-positive breast cancer: pooled analysis of individual patient data from four prospective, neoadjuvant clinical trials. Lancet Oncol. 2021 Aug;22(8):1151-1161. doi: 10.1016/S1470-2045(21)00301-6. Epub 2021 Jul 9. PMID 34252375